CLINICAL TRIAL: NCT05847634
Title: Depth of Sedation and Its Impact on Cerebrovascular Reactivity in Acute Respiratory Distress Syndrome: a Pilot Analysis
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Asher Mendelson, Assistant Professor, University of Manitoba
Other Study IDs: HS25505
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: ARDS, Human
Keywords: Near-Infrared Spectroscopy; Depth of Sedation; Intensive Care Unit; Electroencephalography; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Respiratory Distress Syndrome: Adults admitted to ICU with ARDS confirmed according to Berlin Definition
  Interventions: Device: Masimo O3 NIRS cerebral oximetry and SedLine processed EEG

INTERVENTIONS:
Device: Masimo O3 NIRS cerebral oximetry and SedLine processed EEG — Non-invasive neuromonitoring device for observational study

SUMMARY:
Investigation of the feasibility of monitoring processed transcutaneous electroencephalography (EEG), a method of interpreting brain activity, and near-infrared spectroscopy (NIRS), a method of determining levels of tissue oxygenation (StO2) in the brain, for patients with acute respiratory distress syndrome (ARDS) in the ICU.

DETAILED DESCRIPTION:
The aim of this study is to determine the feasibility of using Masimo SedLine processed EEG monitoring and Masimo O3 NIRS to monitor optimal depth of sedation for patients with ARDS in the ICU.

To achieve this, non-invasive devices will be applied to the participant to measure processed EEG signal and StO2. Cerebrovascular reactivity will be determined using the following two values:

1. SEDopt: The optimal depth of sedation that minimizes correlation between StO2 and processed EEG monitoring.
2. MAPopt: The optimal blood pressure that minimizes correlation between StO2 and MAP.

Demographic information (age, sex, height, weight), past medical history, etiology of ARDS, Disease severity, routine bloodwork, and dose of sedation will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to the ICU
* ARDS confirmed according to the Berlin Definition
* Invasive mechanical ventilation
* Deep sedation and/or neuromuscular blockade required for ARDS treatment at the discretion of the treating medical team
* Application of monitoring devices feasible

Exclusion Criteria:

* More than 24 hours elapsed since ICU admission
* Death is deemed imminent and inevitable during the next 24 hours
* Known allergy to a textile component of the device
* Consent declined from patient or authorized third party
* The treating clinician believes that participation in the study would not be in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the ICU with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 20 months
  Recruitment of two patients per month, allowing for seasonal variation in ARDS.
Data Quality | 7 days
  Physiologic signal with greater than 80% data quality to allow for calculation of SEDopt

SECONDARY OUTCOMES:
SEDopt | 7 days
  Optimal depth of sedation that minimizes correlation between tissue oxygenation (StO2) and total hemoglobin (THb) as measure by O3 NIRS and processed EEG monitoring as defined by SedLine PSi.
MAPopt | 7 days
  Optimal depth of sedation that minimizes correlation between tissue oxygenation (StO2) and mean arterial pressure as measured by invasive arterial line.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Mendelson, MD PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Winnipeg, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No